CLINICAL TRIAL: NCT06375109
Title: PD-L1/PD-1 Inhibitors Plus Chemotherapy Versus Chemotherapy Alone for the Neoadjuvant Treatment of Limited-stage Small Cell Lung Cancer: an Open-label, Non-randomized Controlled, Phase II, Single-center Study
Brief Title: PD-L1/PD-1 Inhibitors Plus Chemotherapy Versus Chemotherapy Alone for the Neoadjuvant Treatment of Limited-stage SCLC
Acronym: NeoSCLC-001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Liang Shi, MD, MD，Associate Chief Physician, Beijing Chest Hospital, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJXK-2023-KY-53; NeoSCLC-001 (Other: Beijing Chest Hospital, Capital Medical University)
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Limited-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tislelizumab; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoCIT (Experimental): Neoadjuvant chemotherapy + Tislelizumab(2-3 cycles), Adjuvant chemotherapy + Tislelizumab (1-2 cycles), Maintenance Tislelizumab
  Interventions: Drug: Tislelizumab; Drug: Carboplatin injection; Drug: Cisplatin injection; Drug: Etoposide injection
- neoCT (Active Comparator): Neoadjuvant chemotherapy (2-3 cycles), Adjuvant chemotherapy (1-2 cycles)
  Interventions: Drug: Carboplatin injection; Drug: Cisplatin injection; Drug: Etoposide injection

INTERVENTIONS:
Drug: Tislelizumab — administered via Intravenous (IV) injection
  Arms: neoCIT
Drug: Carboplatin injection — administered via IV injection
Drug: Cisplatin injection — administered via IV injection
Drug: Etoposide injection — administered via IV injection

SUMMARY:
This is an open-label, non-randomized, controlled, single-center, phase II study to compare the efficacy and safety of neoadjuvant PD-L1/PD-1 inhibitor + chemotherapy (carboplatin/cisplatin + etoposide) with chemotherapy (carboplatin/cisplatin + etoposide) alone followed by radical surgery and adjuvant treatment as perioperative therapy in patients with limited-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in this study, signed an informed consent form, and demonstrated good compliance.
2. They were histologically or cytologically confirmed with limited-stage small-cell lung cancer (TNM stage; T1-3N0-2M0).
3. The age range was 18 to 75 years, with no gender restriction.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score: 0-2.
5. Life expectancy was estimated to be at least 3 months.
6. No previous anti-tumor treatment specifically for SCLC was administered.
7. According to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, there must be at least one measurable lesion.
8. Patients' organ functions must be adequately sufficient, with the following requirements to be met before the first study treatment:

   1. Hematological parameters: ANC ≥1.5×10^9/L, platelets ≥100×10^9/L, hemoglobin ≥90g/L.
   2. Renal function: serum creatinine ≤1.5 times the upper limit, or creatinine clearance ≥50 mL/min.
   3. Liver function: ALT/AST ≤2.5 times the upper limit, total serum bilirubin ≤2 times the upper limit.
   4. Coagulation: INR should be ≤ 1.5 times the upper limit.
9. Patients of childbearing potential must agree to use contraception.
10. Patients must be able to tolerate chemotherapy, immunotherapy, and surgery.

Exclusion Criteria:

1. Patients who have received anti-tumor treatment for SCLC (including but not limited to chemotherapy and radiation therapy at the site of the lesion).
2. Patients who have previously used immune checkpoint inhibitors such as PD-1/PD-L1 inhibitors for treatment.
3. Patients with a history of interstitial lung disease, non-infectious pneumonia, or uncontrollable systemic diseases, including pulmonary fibrosis and acute lung disease.
4. Patients requiring systemic anti-bacterial, anti-fungal, or anti-viral treatment for severe chronic or active infections, including tuberculosis.
5. Patients known to have HIV.
6. Patients with active hepatitis B or hepatitis C.
7. Patients with active autoimmune diseases or a history of autoimmune diseases that may recur.
8. Patients with diseases requiring systemic corticosteroid treatment or other immunosuppressive therapy.
9. Patients deemed by the investigator to have concomitant diseases that pose a serious risk to patient safety or could affect the patient's ability to complete the study.
10. Patients who have undergone major surgery within 4 weeks prior to treatment initiation, or those with significant trauma or fractures, or those with unhealed wounds at the time of treatment.
11. Patients with severe cardiac diseases, such as NYHA class III or higher congestive heart failure, CCS class III or higher angina, a history of myocardial infarction in the past 6 months, or arrhythmias requiring medication.
12. Patients with comorbidities that make them unsuitable for surgery.
13. Patients who have had an allergic reaction to the study drug or excipients in the medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-16 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Up to 3 months following completion of neoadjuvant treatment
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Major Pathologic Response (MPR) Rate | Up to 3 months following completion of neoadjuvant treatment
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy.
Event-Free Survival (EFS) | up to 5 years
  EFS is defined as the time from enrollment until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.
Overall Survival (OS) | up to 5 years
  OS is defined as the time from enrollment until death from any cause.
Objective response rate (ORR) | Up to 1 months following completion of neoadjuvant treatment
  The proportion of patients who have had a complete response or partial response (according to RECIST1.1) in all patients who have completed the neoadjuvant therapy.
  Only patients with measurable lesions at baseline will be analyzed.
Safety: frequency of severe adverse events | up to 6 months
  The frequency of severe adverse events from the participants enrolling to 90 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published